CLINICAL TRIAL: NCT01648218
Title: Insulin Therapy for Post-transplant Glucocorticoid Induced Hyperglycemia
Acronym: PTHG
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, David E. Harris, MD, MD, FRCPC, Clinical Endocrinology Fellow, University of British Columbia, Vancouver General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTHG.VGH.UBC
Record Dates: First submitted 2012-07-12; First posted 2012-07-24 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Post-Transplant Glucocorticoid Induced Diabetes
Keywords: glucocorticoid; diabetes mellitus; post-transplant; insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Insulin; Isophane Insulin, Human; Insulin Aspart; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neutral protamine hagedorn (NPH) insulin (Active Comparator): Drug: Neutral protamine hagedorn (NPH) insulin
  Other Names:
  Humulin N, Novolin N
  Route: Subcutaneous; Dosage: No fixed dose, varies between subjects; Frequency: daily before breakfast; Duration: 12 hours; for duration subjects are concurrently administered once-daily glucocorticoid.
  Interventions: Drug: Neutral protamine hagedorn (NPH) insulin
- Regular or Aspart insulin (Experimental): Drug: Regular human insulin or Insulin Aspart
  Other Names:
  Humulin R, Novolin R, Novolog, NovoRapid
  Route: Subcutaneous; Dosage: No fixed dose, varies between subjects; Frequency: daily before meals; Duration: 2 hours (Aspart) or 6 hours (Regular); for duration subjects are concurrently administered once-daily glucocorticoid.
  Interventions: Drug: Regular human insulin or Insulin Aspart
- Insulin glargine (Experimental): Drug: Insulin glargine
  Other Names:
  Lantus
  Route: Subcutaneous; Dosage: No fixed dose, varies between subjects; Frequency: daily before breakfast; Duration: 24 hours; for duration subjects are concurrently administered once-daily glucocorticoid.
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: Neutral protamine hagedorn (NPH) insulin
  Other Names: Humulin N, Novolin N
  Arms: Neutral protamine hagedorn (NPH) insulin
Drug: Regular human insulin or Insulin Aspart
  Other Names: Humulin R; Novolin R; Novolog; NovoRapid
  Arms: Regular or Aspart insulin
Drug: Insulin glargine
  Other Names: Lantus
  Arms: Insulin glargine

SUMMARY:
No consensus guidelines exist for management of post-transplant glucocorticoid induced hyperglycemia, but most published reviews recommend insulin as first line therapy. A variety of insulin regimens have been proposed, including mealtime short-acting regular or analog insulin, once daily neutral protamine hagedorn (NPH) insulin, pre-mixed insulin, or basal insulin alone such as glargine or detemir. However, no randomized trial has ever examined different insulin regimens to determine which most effectively controls post-transplant steroid-induced hyperglycemia. Consequently, the proposed study intends to examine three commonly used insulin regimens used for managing post-transplant once-daily glucocorticoid-induced hyperglycemia to determine which is most effective:

* Group 1: Intermediate-acting (NPH) insulin at breakfast
* Group 2: Short-acting insulin (regular or aspart) before meals
* Group 3: Insulin glargine at breakfast

Question/Hypothesis:

Among three commonly used insulin regimens, which is most effective for managing post-transplant once-daily glucocorticoid-induced hyperglycemia?

ELIGIBILITY:
Inclusion Criteria:

1. Have undergone bone marrow, liver, lung, or renal transplant.
2. Be using once daily oral glucocorticoid therapy (total daily dose of Prednisone ≥10 mg, Hydrocortisone ≥40 mg, Dexamethasone ≥1.5 mg) administered in the morning and expected to continue for at least 2 weeks.
3. Have pre-existing or newly diagnosed diabetes mellitus established by any of the criteria listed below:

   1. Fasting plasma glucose ≥7.0 mmol/L (repeated x 1)
   2. Any plasma glucose ≥11.0 mmol/L
4. Have at least three pre-meal inpatient capillary blood glucose (CBG) readings ≥ 7.8 mmol/L
5. Be eating meals by mouth

Exclusion Criteria:

1. Heart, Pancreas, Islet cell transplant recipients
2. Previous use of Basal-Bolus or Pre-Mixed Insulin regimen
3. Diabetes mellitus type I
4. NPO (not eating meals by mouth)
5. Receiving enteral (tube feeds) or parenteral (TPN) nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Blood glucose - inpatient | Time (days) from enrollment to described treatment range, an expected average of 7 days
  Mean time from baseline to achieve at least 80% of pre-meal capillary blood glucose values within 5.0 - 7.8 mmol/L over a 48 hour period during hospitalization

SECONDARY OUTCOMES:
Blood glucose - inpatient | Subjects will be followed from enrollment for the remainder of hospital stay (days), an expected average of 21 days
  Mean inpatient capillary blood glucose (mmol/L) from enrollment to discharge from hospital
Post prandial blood glucose - inpatient | Subjects will be followed from enrollment for the remainder of hospital stay (days), an expected average of 21 days
  Mean inpatient two-hour post-lunch capillary blood glucose (mmol/L) from enrollment to discharge from hospital
Length of inpatient hospital stay | Subjects will be followed from enrollment for the remainder of hospital stay (days), an expected average of 21 days
  Length of stay in hospital (days) from enrollment to discharge from hospital
Blood glucose | Enrollment to 3 months
  Mean fasting blood glucose (mmol/L) from enrollment to 3 months
Hemoglobin A1C | Enrollment to 3 months
  Mean hemoglobin A1C (%) from enrollment to 3 months
Post prandial blood glucose | Enrollment to 3 months
  Mean two-hour post-lunch capillary blood glucose (mmol/L) from enrollment to 3 months
Hypoglycemic episodes | Enrollment to 3 months
  Hypoglycemic episodes defined as:
  (1) Mild - any measured CBG 3.0-4.0 mmol/L; (2) Severe - any episode of hypoglycemia with a measured CBG < 3.0 mmol/L, OR which the subject is not able to recognize and treat without the direct (substantial) intervention of a professional caregiver, nurse or physician (e.g. intravenous dextrose or intramuscular glucagon)
Glycemic treatment failure | Enrollment to 3 months
  Hypoglycemic treatment failure: subject experiences ≥3 hypoglycemic episodes (≤ 4.0 mmol/L) over any 5 day period or a single severe hypoglycemic event (as previously defined), they will be withdrawn from study and managed at discretion of attending physician, or hospital endocrine consult service.
  Hyperglycemic treatment failure: Severe hyperglycemia defined as CBG >20 mmol/L. If subject experiences ≥3 severe hyperglycemic measures over the course of 48 hours they will be withdrawn from the study and managed at discretion of attending physician, or hospital endocrine consult service.
Cardiovascular events | Enrollment to 3 months
  New cardiovascular events defined as: myocardial infarction, new or worsened congestive heart failure, stroke, and cardiac arrhythmia.
Post-transplant infections or new antibiotic use | Enrollment to 3 months
  Post-transplant infections or new antibiotic use from enrollment to 3 months.
Transplant graft failure | Enrollment to 3 months
  Transplant graft failure (as specified by subject's medical transplant physician) from enrollment to 3 months.
New acute renal failure | Enrollment to 3 months
  New acute renal failure is defined according to Acute Kidney Network Guidelines: rapid time course and decreased kidney function according to an absolute Creatinine (Cr) rise greater than 26 μmol/L, greater than 2-fold increase in serum Cr from baseline, or urine output less than 0.5 mL/kg/hr for greater than 6 hours
Mortality | Enrollment to 3 months
  Overall subject mortality from baseline to 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Breay W Paty, MD, FRCPC, Principal Investigator — Vancouver General Hospital, University of British Columbia
Locations (1):
- Vancouver General Hospital - Jim Pattison Pavilion, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Lane JT, Dagogo-Jack S. Approach to the patient with new-onset diabetes after transplant (NODAT). J Clin Endocrinol Metab. 2011 Nov;96(11):3289-97. doi: 10.1210/jc.2011-0657. PMID 22058376
- [Background] Sarno G, Muscogiuri G, De Rosa P. New-onset diabetes after kidney transplantation: prevalence, risk factors, and management. Transplantation. 2012 Jun 27;93(12):1189-95. doi: 10.1097/TP.0b013e31824db97d. PMID 22475764
- [Background] Griffith ML, Jagasia M, Jagasia SM. Diabetes mellitus after hematopoietic stem cell transplantation. Endocr Pract. 2010 Jul-Aug;16(4):699-706. doi: 10.4158/EP10027.RA. PMID 20439241
- [Background] Lansang MC, Hustak LK. Glucocorticoid-induced diabetes and adrenal suppression: how to detect and manage them. Cleve Clin J Med. 2011 Nov;78(11):748-56. doi: 10.3949/ccjm.78a.10180. PMID 22049542
- [Background] Umpierrez GE, Hellman R, Korytkowski MT, Kosiborod M, Maynard GA, Montori VM, Seley JJ, Van den Berghe G; Endocrine Society. Management of hyperglycemia in hospitalized patients in non-critical care setting: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2012 Jan;97(1):16-38. doi: 10.1210/jc.2011-2098. PMID 22223765
- See also: Multilingual dietary instructions to be distributed to ALL subjects during study from the Canadian Diabetes Association — http://www.diabetes.ca/diabetes-and-you/nutrition/just-basics/